CLINICAL TRIAL: NCT01780688
Title: A Single-center, Open-label, Randomized, Controlled, Crossover Study to Explore the Nicotine Pharmacokinetic Profile and Safety of Tobacco Heating System (THS) 2.1 Compared to Conventional Cigarettes Following Single and ad Libitum Use in Smoking, But Otherwise Healthy Subjects.
Brief Title: Exploratory THS 2.1 Nicotine Pharmacokinetics and Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZRHX-PK-02
Record Dates: First submitted 2013-01-15; First posted 2013-01-31 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Smoking
Keywords: Modified risk tobacco product (MRTP); Smoking; Nicotine profile
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- smoking conventional cigarettes (CC) (Active Comparator): After a 1-day nicotine deprivation, subjects are smoking one single cigarette (usual own brand) on one day and then smoking ad libitum on the subsequent day
  Interventions: Other: Conventional cigarettes (CC); Other: THS 2.1
- using the Tobacco Heating System 2.1 (THS 2.1) (Experimental): After a 1-day nicotine deprivation, subjects are puffing one single tobacco stick using the THS 2.1 on one day and then puffing ad libitum on the subsequent day
  Interventions: Other: Conventional cigarettes (CC); Other: THS 2.1

INTERVENTIONS:
Other: Conventional cigarettes (CC) — Subjects are randomized in a 1:1 fashion to be assigned to one of the 2 sequences, either A) CC and then THS 2.1, or B) THS 2.1 and then CC.
Other: THS 2.1 — Subjects are randomized in a 1:1 fashion to be assigned in one of the sequences, either A) CC and then THS 2.1, or B) THS 2.1 and then CC

SUMMARY:
The main goal of this exploratory study is to evaluate the pharmacokinetic profile of nicotine for the candidate modified risk tobacco product THS 2.1 and for conventional cigarettes (CC).

DETAILED DESCRIPTION:
This 2-period 2-sequence cross-over clinical study intends to explore the profile of nicotine uptake (rate and extent of nicotine absorbed and associated variability) in healthy smokers switching from (CC) to THS 2.1 (single or ad libitum use) compared to smokers continuing to use CC, as a comparator. This study will serve to optimize blood sampling schedules and sample size estimation for further studies. This study will also provide preliminary information on the relationship between nicotine absorption and urge to smoke/withdrawal symptoms when using THS 2.1 as compared to CC, as well as the safety profile, which is related to the use of THS 2.1.

After screening, enrolled subjects will be admitted to the clinic for 8 days. This study duration includes 2 consecutive periods. Each period consists of 1 day for single use of the product preceded by a 24-hour nicotine deprivation, and 1 day for ad libitum product use. After leaving the clinic, the subjects will be followed up for safety over a period of 7 days.

This clinical study will be conducted in compliance with International Conference on Harmonisation of technical requirements for registration of pharmaceuticals for human use (ICH Good Clinical Practice), the Declaration of Helsinki as amended in 2008, and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed an informed consent form before commencement of study procedures
* Healthy Caucasian aged between 23 to 65 years
* Subject is current smoker for at least 3 years (based on self-reporting and biochemically verified), who, for the last 4 weeks, had smoked at least 10 commercially available non-mentholated CC per day, and is not planning to make a quit attempt within the next 3 months

Exclusion Criteria:

* As per Investigator judgment, the subject should not participate in the study for any reason (e.g. medical, psychiatric and/or social reason)
* The subject has a medical condition requiring smoking cessation, or has a clinically relevant disease / condition which could interfere with the study participation and/or study results
* The subject has participated in a clinical study within 3 months prior to the Screening Visit
* Pregnant or lactating woman, and for woman of childbearing potential, absence / refusal to use an acceptable method of effective contraception

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Nicotine Cmax | Single use (1 day)
  Maximum plasma concentration (Cmax)
Nicotine AUC | Single use (1 day)
  Nicotine plasma concentration, area under the curve (AUCt)

SECONDARY OUTCOMES:
Nicotine concentrations | Single use (1 day); multiple use (1 day)
  Time course of plasma nicotine concentration
Questionnaire of smoking urges (brief version) (QSU-brief) | single use (1 day); multiple use (1 day)
  QSU-brief measuring subjective effects of smoking
Safety monitoring | 7 days + 7 days follow-up
  Monitoring of adverse events, based on clinical and laboratory evaluation
Nicotine tmax | Single use (1 day)
  Time to maximal nicotine concentration in plasma
Cough Visual Analog Scale | 7 days
  Visual Analog Scale on cough
Modified Cigarette Evaluation Questionnaire (MCEQ) | single use (1 day); multiple use (1 day)
  MCEQ measuring effects of smoking

CONTACTS AND LOCATIONS:
Overall Officials: Adrian J Stewart, MD, Principal Investigator — Celerion, Belfast, Northern Ireland
Locations (1):
- Celerion, 22-24 Lisburn Road, Belfast, United Kingdom

REFERENCES:
- [Result] Picavet P, Haziza C, Lama N, Weitkunat R, Ludicke F. Comparison of the Pharmacokinetics of Nicotine Following Single and Ad Libitum Use of a Tobacco Heating System or Combustible Cigarettes. Nicotine Tob Res. 2016 May;18(5):557-63. doi: 10.1093/ntr/ntv220. Epub 2015 Oct 5. PMID 26438645